CLINICAL TRIAL: NCT06679517
Title: Studio OsseRvaziOnAle RelatIvo Al Follow-up a LuNGo Termine Di Pazienti Con Stenosi Aortica Severa Valutati Per Sostituzione Valvolare Aortica Percutanea (TAVI).
Brief Title: Observational Study Relating to the Long-term Follow-up of Patients with Severe Aortic Stenosis Evaluated for Percutaneous Aortic Valve Replacement (TAVI).
Acronym: ROARING-TAVI
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Rita Pavasini, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 519/2024/Oss/AOUFe
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Severe Aortic Stenosis; TAVI(Transcatheter Aortic Valve Implantation)
Keywords: severe aortic stenosis; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with aortic stenosis undergoing TAVI: Patients with a diagnosis of severe aortic stenosis candidates to TAVI procedures.
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI — Clinical follow-up up to 10 years of patients undergoing TAVI

SUMMARY:
All patients with severe aortic stenosis undergoing evaluation for TAVI are routinely subjected to a series of assessments:

* Pre-implantation: thoraco-abdominal CT angiography, coronary angiography, echocardiography, clinical assessment, ECG, and laboratory tests.
* Post-implantation: echocardiography, laboratory tests, ECG, assessment of any procedural complications, and a cardiology follow-up visit.

This is an observational study, with the aim to monitor over time the population of patients who have undergone TAVI, identifying pre- and post-implant conditions that may negatively impact patient outcomes (both clinical factors and those directly related to the prosthetic implant). Through a 10-year follow-up, the study seeks to determine the incidence of prosthetic failure, as well as the incidence of prosthesis-related complications and major clinical endpoints.

DETAILED DESCRIPTION:
DESIGN OF THE STUDY

This is a retrospective and prospective observational, non-profit study. All consecutive patients who have entered the TAVI pathway at this hospital (Azienda Ospedaliera Universitaria di Ferrara) since January 2016 will be included in the study.

The study does not involve any alteration or modification of routine clinical practice and does not require any center or operator to use specific devices.

It involves the collection of pre- and post-procedural data from patients who enter the TAVI pathway.

All patients will be re-contacted to confirm clinical follow-up via telephone to gather information on any adverse events that may have occurred in the years following TAVI (at 1, 5, and 10 years post-TAVI).

For each patient enrolled in the study, an anonymous case report form (CRF) will be completed.

INCLUSION AND EXCLUSION CRITERIA

All patients referred to the valve disease outpatient clinic with a diagnosis of severe aortic stenosis who are candidates for TAVI will be asked to participate in the study and sign the consent form as part of the process to schedule the required investigations.

All consecutive patients with a diagnosis of severe aortic stenosis who, since January 2016, who have completed all the clinical and instrumental investigations required by the hospital protocol prior to receiving TAVI will be enrolled. Therefore, all patients with a diagnosis of severe aortic stenosis who have been indicated for TAVI and have completed the following will be included in the study:

1. Pre-TAVI transthoracic echocardiogram
2. ECG and cardiology consultation to confirm TAVI eligibility
3. Thoraco-abdominal aortic CT angiography
4. Coronary angiography +/- angioplasty +/- valvuloplasty. The decision to perform valvuloplasty or angioplasty prior to TAVI remains at the discretion of the operating physician.

This protocol does not alter clinical judgment or daily routine in any way.

Inclusion criteria:

Age >18 years Signing of the consent form Diagnosis of severe aortic stenosis with an indication for TAVI Completion of the required TAVI pathway exams (ECG and cardiology consultation, echocardiogram, thoraco-abdominal aortic CT angiography, coronary angiography)

Exclusion criteria:

Lack of signed consent form Inability to complete follow-up

CONSENT ACQUISITION AND STUDY ENROLLMENT

When a patient meeting the inclusion and exclusion criteria is identified, the investigator or their delegate will explain the study, its procedures, and objectives to the patient. If the patient agrees to participate, they must sign the consent form. The investigator is responsible for keeping a copy of the consent form and providing one to the patient. After consent is signed, all baseline patient characteristics and procedural details will be documented in the designated CRF.

In line with current recommendations for clinical study management, a unique identifier will be assigned to each patient upon creation of the CRF to ensure traceability. Only the investigator will be able to link this identifier to the patient for follow-up purposes. No one other than the center's investigator will have access to identifying patient information in the CRF.

The study also includes a retrospective component, for which patient data will be used in anonymized form. In the retrospective phase, consent will also be obtained for data use, except in cases where patients are deceased or unreachable. In the former case, consent from family members will be sought, while in the latter, the patient will not be included in the study.

The Principal Investigator (PI) or their delegate will collect the following information for each enrolled patient, which will be recorded in the CRF. Documentation of adverse events should be as thorough as possible to enable assessment by the independent adverse event adjudication committee.

ASSESSMENTS PERFORMED IN THE TAVI PATHWAY

As part of standard clinical practice, all patients entering the TAVI pathway will undergo the following:

* Electrocardiogram and cardiology consultation
* Complete transthoracic echocardiogram
* Thoraco-abdominal CT angiography
* Coronary angiography +/- angioplasty +/- valvuloplasty

PROSTHESIS IMPLANTATION INFORMATION

During the TAVI hospitalization, the following clinical information will be collected for each enrolled patient:

Type of implanted prosthesis Procedural details (fluoroscopy time, amount of contrast media, use of temporary pacemaker) Information on any procedural or post-procedural complications according to VARC criteria (see subsequent definitions) POST-TAVI ASSESSMENTS

Following TAVI, as per routine practice, patients will undergo the following evaluations before discharge (at our hospital in case of in-service procedures or at the TAVI-performing center):

Electrocardiogram Transthoracic echocardiogram Clinical assessment to rule out post-procedural complications

CLINICAL FOLLOW-UP

All TAVI patients are routinely re-evaluated 1-3 months post-procedure at the Valve Disease outpatient clinic, where they receive:

Clinical assessment Electrocardiogram Transthoracic echocardiogram

TELEPHONE FOLLOW-UP All patients enrolled in the study will be contacted by telephone at 1, 5, and 10 years post-TAVI to gather information on any adverse events that may have occurred during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years Signing of the consent form Diagnosis of severe aortic stenosis with an indication for TAVI Completion of the required TAVI pathway exams (ECG and cardiology consultation, echocardiogram, thoraco-abdominal aortic CT angiography, coronary angiography)

Exclusion Criteria:

Lack of signed consent form Inability to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with a diagnosis of severe aortic stenosis who, since January 2016, have completed all the clinical and instrumental investigations required by the hospital protocol prior to receiving TAVI will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2035-11-30 (Estimated); Study Completion 2035-11-30 (Estimated)

PRIMARY OUTCOMES:
Prosthesis failure | 10 years
  Valve-related mortality OR aortic valve reintervention OR Stage III hemodynamic valve deterioration.

SECONDARY OUTCOMES:
composite of all-cause death, stroke and myocardial infarction | 1, 5 and 10 years
  composite of all-cause death, stroke and myocardial infarction
all-cause death | 1, 5 and 10 years
  all-cause death
myocardial infarction | 1, 5 and 10 years
  myocardial infarction
stroke or transient ischemic attack | 1, 5 and 10 years
  Any new cerebrovascular accident
atrial fibrillation | 1, 5, 10 years
  new onset atrial fibrillation
pacemaker implantation | 1, 5 and 10 years
  pacemaker implantation after the TAVI procedure
endocarditis | 1, 5 and 10 years
  endocarditis of the TAVI
re-hospitalization | 1,5 and 10 years
  new all-cause hospitalization after TAVI
prosthesis failure | 1 and 5 years
  Valve-related mortality OR aortic valve reintervention OR Stage III hemodynamic valve deterioration.
single component of the primary endpoint | 10 years
  Valve-related mortality OR aortic valve reintervention OR Stage III hemodynamic valve deterioration.
incidentalomas | 1, 5 and 10 years
  rate of incidentalomas at the TAVI pre-screening exams
prosthesis failure in patients with incidentaloma | 1 and 5 years
  occurrence of prothesis failure in patients with incidentaloma
re-TAVI or SVAR in TAVI | 5 and 10 years
  Occurence of re-intervention with TAVI or surgically in patients treated with TAVI
coronary revascularization | 1 and 5 years
  new coronary revascularization after TAVI
complication after valvuloplasty pre-TAVI | in-hospital, 1 year
  occurrence of any complication following aortic valvuloplasty pre-TAVI
CT predictors of complications post valvuloplasty | 1 year
  Presence of predictors of complications related to valvuloplasty on CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided